CLINICAL TRIAL: NCT03744585
Title: Cabozantinib Real-life Use for Advanced Renal Cell Carcinoma in France: a Retrospective Descriptive Non-interventional Study of 2 Cohorts.
Acronym: CABOREAL
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-FR-60000-006
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Subjects who received at least one dose of cabozantinib during the Authorization for Use (ATU) period (12/09/2016 to 09/12/2016) for the treatment of advanced Renal Cell Carcinoma (RCC).
- Cohort 2: Subjects who received at least one dose of cabozantinib during the first six months after the ATU period (10/12/2016 to 16/02/2018).

SUMMARY:
The primary objective of the study is to describe the real-life conditions of use and exposure of cabozantinib in France in two cohorts defined by their treatment initiation period.

ELIGIBILITY:
Inclusion Criteria:

* Any subjects from the participating sites (dead or alive) who have received at least one dose of cabozantinib within the ATU program or between 10/12/2016 and 16/02/2018 and for whom the medical file is available

Exclusion Criteria:

* Patients alive at study initiation who have not received information notice
* who have opposed to data collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort 1: subjects who received at least one dose of cabozantinib during the ATU period (12/09/2016 to 09/12/2016) for the treatment of advanced RCC. Cohort 2: subjects who received at least one dose of cabozantinib during the first six months after the ATU period (10/12/2016 to 16/02/2018).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Duration of treatment exposure | during the whole study period for a maximum of 28 to 31 months
Dose prescribed at initiation | during the whole study period for a maximum of 28 to 31 months
Average Daily Dose | during the whole study period for a maximum of 28 to 31 months
  average daily dose received by subject during the treatment exposure
Number of subjects with ≥1 temporary interruptions | during the whole study period for a maximum of 28 to 31 months
Number of interruptions per subject | during the whole study period for a maximum of 28 to 31 months
Number of subjects with ≥1 dose modification(s) | during the whole study period for a maximum of 28 to 31 months
Number of subjects with permanent discontinuations | during the whole study period for a maximum of 28 to 31 months

SECONDARY OUTCOMES:
Overall survival of subjects since cabozantinib initiation | during the whole study period for a maximum of 28 to 31 months
Overall survival of subjects since RCC diagnosis. | during the whole study period for a maximum of 28 to 31 months
Overall survival of subjects since metastatic diagnosis | during the whole study period for a maximum of 28 to 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France

REFERENCES:
- [Derived] Albiges L, Flechon A, Chevreau C, Topart D, Gravis G, Oudard S, Tourani JM, Geoffrois L, Meriaux E, Thiery-Vuillemin A, Barthelemy P, Ladoire S, Laguerre B, Perrot V, Billard A, Escudier B, Gross-Goupil M. Real-world evidence of cabozantinib in patients with metastatic renal cell carcinoma: Results from the CABOREAL Early Access Program. Eur J Cancer. 2021 Jan;142:102-111. doi: 10.1016/j.ejca.2020.09.030. Epub 2020 Nov 27. PMID 33253997